CLINICAL TRIAL: NCT02688868
Title: The Safety and Effectiveness Evaluation of New Specifications (2.25mm) of FirehawkTM Sirolimus Target-eluting Coronary Stent System in the Treatment of Coronary Heart Disease: a Prospective, Multicenter, Single-group Study.
Brief Title: Evaluation of New Specifications (2.25mm) of FirehawkTM in the Treatment of Coronary Heart Disease ( Firehawk_2.25 )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Firehawk_SS
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2020-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- new specifications (Diameter 2.25mm)of Firehawk stent (Experimental): Evaluation of new specifications (Diameter 2.25mm) of FirehawkTM in the treatment of coronary heart disease
  Interventions: Device: FirehawkTM 2.25mm

INTERVENTIONS:
Device: FirehawkTM 2.25mm — Implantation of the released specification (2.25mm) of FirehawkTM rapamycin target-eluting coronary stent systems

SUMMARY:
The purpose of this study is to evalute the clinical safety and effectiveness of released specification (2.25mm) of FirehawkTM Sirolimus target-eluting coronary stent system.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age, males or non-pregnant women;
2. Evidence of silent ischemia, stability or in patients with old myocardial infarction or unstable angina;
3. Primary target lesion, in situ coronary artery disease;
4. Target lesion length ≤ 60mm, target lesion diameter 2.25mm (Visual method);
5. The target lesion diameter stenosis ≥ 70% (Visual method);
6. Each target lesion implantation the same stent (Firehawk stent);
7. With indications for coronary artery bypass surgery;
8. To understand the purpose of testing, voluntary and informed consent, patients agreed to achieve invasive imaging and clinical follow-up.

Exclusion Criteria:

1. Within 72h of any acute myocardial infarction;
2. Unprotected left main coronary artery disease, triple vessel lesions which need treated all; bifurcation lesions and vascular lesions of the bridge;
3. Severe calcified lesions that cannot be successfully expanded and distorting lesions not suitable for stent delivery;
4. Artery and/or vein bypass graft lesions;
5. Intracoronary implantation of any branding stents within 1 year;
6. Severe congestive heart failure (NYHA class III and above), or left ventricular ejection fraction <35% (ultrasound or left ventricular angiography);
7. Preoperative renal function serum creatinine >2.0mg/DL;
8. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
9. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
10. The patient's life expectancy is less than 12 months;
11. Top participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
12. Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
13. Heart transplantation patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Principal Investigator — Fu Wai Hospital & National Center for Cardiovascular Diseases in China
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Started | 38
Completed | 34
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.22 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 25
Region of Enrollment [Number; unit: participants]
  China | 38

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Loss
Description: the difference between the minimal lumen diameter immediately after stent implantation and the minimal lumen diameter by angiography review 9 months after the procedure.
Time Frame: 9 month after stent implantation
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 34
mm | 0.29 (0.57)

2. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: including cardiac death, target vessel myocardial infarction and clinical symptom-driven target lesion revascularization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 38
Participants | 3

3. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 38
Participants | 4

4. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 3 years
Population: One missed participant in 3 years follow up
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 37
Participants | 4

5. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 4 years
Population: Two missed participant in 4 years follow up
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 36
Participants | 4

6. Secondary Outcome: Number of Participants With MACE
Description: a composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 38
Participants | 6

7. Secondary Outcome: Number of Participants With MACE
Description: a composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 38
Participants | 10

8. Secondary Outcome: Number of Participants With MACE
Description: a composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 3 years
Population: One missed participant in 3 years follow up
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 37
Participants | 10

9. Secondary Outcome: Number of Participants With MACE
Description: a composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 4 years
Population: One missed participant in 3 years follow up
Measure: Count of Participants; unit: Participants
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
Number analyzed (Participants) | 37
Participants | 11

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | New Specifications (Diameter 2.25mm)of Firehawk Stent
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 28/38
Other Adverse Events (participants affected / at risk) | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Specifications (Diameter 2.25mm)of Firehawk Stent (N=38)
target lesion revascularization (Cardiac disorders) | 3 (3)
in-stent restenosis (Cardiac disorders) | 1 (1)
angina (Cardiac disorders) | 2 (2)
hypotension (Vascular disorders) | 1 (1)
rehospitalization (General disorders) | 10 (10)
non target lesion revascularization (Cardiac disorders) | 6 (6)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
renal artery implantation (Vascular disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
Death of cerebral infarction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Specifications (Diameter 2.25mm)of Firehawk Stent (N=38)
elevated myocardial enzyme (Cardiac disorders) | 5 (5)
No-reflow phenomenon (Cardiac disorders) | 1 (1)
intermediate lesion (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Repeat chest & back pain (General disorders) | 3 (3)
atrial fibrillation (Cardiac disorders) | 1 (1)
abnormal liver function (General disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spondylopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
soft tissue disease (Skin and subcutaneous tissue disorders) | 1 (1)
perioperation hypotension (Vascular disorders) | 1 (1)
perioperation slow heart beat (Cardiac disorders) | 1 (1)
Sleeping disorder (Psychiatric disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
Gastroesophageal disorder (Gastrointestinal disorders) | 1 (1)
Varicosity (Vascular disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Heart dysfunction (Cardiac disorders) | 1 (1)
Myocardial injury (Cardiac disorders) | 10 (10)
rapid heart beat (Cardiac disorders) | 1 (1)
Chest distress (Cardiac disorders) | 5 (5)
Chest pain (Cardiac disorders) | 6 (6)
unsatifactory blood glucose control (Metabolism and nutrition disorders) | 1 (1)
lumbago (Skin and subcutaneous tissue disorders) | 1 (1)
Deaf (Ear and labyrinth disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
peripheral neuropathy (Nervous system disorders) | 1 (1)
disc herniation (Nervous system disorders) | 1 (1)
Fasciitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes